CLINICAL TRIAL: NCT00003487
Title: Phase II Study of Antineoplastons A10 and AS2-1 In Patients With Adenocarcinoma of the Esophagus
Brief Title: Antineoplaston Therapy in Treating Patients With Cancer of the Esophagus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066525; BC-ES-2 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Adenocarcinoma of the Esophagus
Keywords: esophageal cancer; recurrent esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with Adenocarcinoma of the Esophagus will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
Current therapies for Adenocarcinoma of the Esophagus provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Adenocarcinoma of the Esophagus.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Adenocarcinoma of the Esophagus.

DETAILED DESCRIPTION:
Esophageal cancer patients receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with esophageal cancer, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Esophageal Cancer.
* To determine objective response, tumor size is measured utilizing physical examination, and radiologic studies performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the esophagus that is unlikely to respond to existing therapy and for which no curative therapy exists
* Meets 1 of the following criteria:

  * Metastatic disease
  * Not curable with surgery or radiotherapy
* Measurable disease by MRI or CT scan

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2000/mm3
* Platelet count at least 50,000/mm3

Hepatic:

* No hepatic failure
* Bilirubin no greater than 2.5 mg/dL
* SGOT and SGPT no greater than 5 times upper limit of normal

Renal:

* Creatinine no greater than 2.5 mg/ml
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No chronic or congestive heart failure
* No uncontrolled hypertension
* No other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No serious lung disease, such as severe chronic obstructive pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No medical illness, psychiatric illness, or non-malignant systemic disease that would preclude study treatment
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered

Endocrine therapy:

* Concurrent steroids allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy (except in patients with multiple tumors who have received radiotherapy to some of their tumors) and recovered

Surgery:

* Recovered from prior surgery

Other:

* No prior antineoplaston therapy
* Prior cytodifferentiating agents allowed

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 1996-05-30 (Actual); Primary Completion 2001-04-27 (Actual); Study Completion 2001-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 8
Completed | 6
Not Completed | 2
Not completed — Not evaluable | 2

BASELINE CHARACTERISTICS:
Population: Eight patients were enrolled in the study, only six were evaluable.
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 52.2 [38.5 to 69.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response, Stable Disease, Progressive Disease or Not Evaluable
Description: Objective response rate per The International Working Group response criteria (1999): Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable lesions, sustained for at least four weeks. Stable Disease (SD), < 50% change in the sum of the products of of the greatest perpendicular diameters of all measurable lesions, sustained for at least twelve weeks.
Time Frame: 59 months
Population: All patients enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 8
participants | 8

ADVERSE EVENTS:
Time Frame: 4 years, 11 months
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 5/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=8)
Hemoglobin (Blood and lymphatic system disorders) | 1
Hypotension (Cardiac disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Hemorrhage: Gastrointestinal (Gastrointestinal disorders) | 4
Infection: Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=8)
Allergic reaction/hypersensitivity (including drug fever) (General disorders) | 1
Hearing (without monitoring program) (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 6
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2
Hypertension (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Non-functional Central Venous Catheter (General disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4
Fever (General disorders) | 4
Rigors/chills (General disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Edema/Fluid retention (General disorders) | 4
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 4
Hemorrhage, GI (Gastrointestinal disorders) | 5
Infection (documented clinically): Abdomen NOS (Infections and infestations) | 1
Infection (documented clinically): Blood (Infections and infestations) | 1
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 2
Infection (documented clinically): Small bowel NOS (Infections and infestations) | 1
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 3
Opportunistic infection (Infections and infestations) | 4
Albumin, serum-low (hypoalbuminemia) (Investigations) | 3
Alkaline phosphatase (Investigations) | 3
Hyperbilirubinemia (Investigations) | 1
Hyperglycemia (Investigations) | 5
Hyperkalemia (Investigations) | 1
Hypernatremia (Investigations) | 4
Hypocalcemia (Investigations) | 5
Hypoglycemia (Investigations) | 2
Hypokalemia (Investigations) | 6
Hypomagnesemia (Investigations) | 1
Metabolic/Laboratory - Other (Investigations) | 1
SGOT (Investigations) | 2
SGPT (Investigations) | 2
Uric acid, serum-high (hyperuricemia) (Investigations) | 2
Confusion (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Somnolence/depressed level of consciousness (Nervous system disorders) | 3
Pain: Back (Musculoskeletal and connective tissue disorders) | 2
Pain: Chest wall (Musculoskeletal and connective tissue disorders) | 1
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 1
Pain: Pain NOS (General disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Flu-like illness (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No